CLINICAL TRIAL: NCT02159833
Title: Phase 1/2 Study to Determine the Intranasal Allergen Threshold to Food Proteins in Children With Food Allergy
Brief Title: Intranasal Diagnostics in Food Allergy: a Feasibility Study
Acronym: INDY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14SM2069
Record Dates: First submitted 2014-06-03; First posted 2014-06-10 (Estimated); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Food Allergy
Keywords: Food allergy; Diagnosis
MeSH Terms: conditions — Food Hypersensitivity; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Intranasal challenge with food protein or vehicle control
  Interventions: Other: Intranasal challenge with active substance (food protein); Other: Intranasal challenge with placebo

INTERVENTIONS:
Other: Intranasal challenge with active substance (food protein)
Other: Intranasal challenge with placebo
  Other Names: placebo = 0.9% NaCl saline solution

SUMMARY:
The investigators will conduct low-dose intranasal allergen challenges on children/adolescents with a diagnosis of food allergy to egg/cow's milk/soya/wheat/peanut. The data will be used to determine the safety and potential utility of intranasal food challenges in the diagnosis of food allergy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 6 - 17 years old
* Physician-diagnosis of food allergy on the basis of:

  * Positive oral food challenge to the causative food (conducted under medical supervision) within the last 12 months; OR
  * History of convincing clinical reaction to the causative food within the last 12 months AND positive skin prick test within last 12 months; OR
  * Evidence of >95% likelihood of food allergy (on the basis of serum specific IgE or skin prick test (SPT) 8mm or above to the causative food allergen within past 12 months
* Written informed consent from parent/guardian, with assent from children aged 8 years and above wherever possible. Participants aged over 16 years will need to provide their owned informed consent.

Exclusion Criteria:

* Contraindicated as acutely unwell or current unstable asthma:

  * Acute wheeze in last 72 hours requiring treatment
  * Febrile ≥38.0oC in last 72 hours
  * Recent admission to hospital in last 2 weeks for acute asthma
* Current medication

  * Use of asthma reliever medication in last 72 hours
  * Recent administration of a medication containing antihistamine within the last 4 days
  * Current oral steroid for asthma exacerbation or course completed within last 2 weeks

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Physiological response to intranasal challenge with a food protein | 20mins
  The physiological response to food (egg/cow's milk/soya/wheat/peanut) protein when administered into the human nasal airway in food-allergic children with the corresponding food allergy. This will be assessed objectively (using acoustic rhinometry and peak nasal inspiratory flow) as well as subjectively (using a validated Symptom Scoring questionnaire).

SECONDARY OUTCOMES:
Intranasal threshold to food protein | 20 mins
  The intranasal threshold to food (egg/cow's milk/soya/wheat/peanut) protein to elicit a local physiological response in food-allergic children (with the corresponding food allergy), as defined by objective assessment described above.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Turner, FRACP PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London / Imperial College Healthcare NHS Trust, London, United Kingdom